CLINICAL TRIAL: NCT00108940
Title: Siblings With Ischemic Stroke Study
Acronym: SWISS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: James F. Meschia, MD, Mayo Clinic College of Medicine Jacksonville
Other Study IDs: 1082-99; R01NS039987 (NIH)
Record Dates: First submitted 2005-04-20; First posted 2005-04-21 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Stroke
Keywords: stroke; ischemic stroke; siblings
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find the genes that increase the risk of developing an ischemic stroke using DNA samples collected from concordant (stroke-affected) sibling pairs.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death in the United States and a leading cause of acquired disability in adults. Each year, about 700,000 people experience stroke in the country. Ischemic stroke, which constitutes about 80 percent of all strokes, is a complex genetic disorder--the result of interactions between multiple genes and multiple environmental exposures. Genes affecting cholesterol, blood pressure, clotting, and other factors may increase the risk of ischemic stroke.

In this clinical study, investigators are studying groups of siblings in which at least two of the siblings have had an ischemic stroke. The goal of this multi-center study is to find the genes that increase the risk of developing an ischemic stroke.

To accomplish the aims of the study, researchers are using DNA samples collected from concordant (stroke-affected) sibling pairs to determine if there are regions in the human genome associated with ischemic stroke or that may harbor stroke susceptibility genes.

Two teaspoons of blood will be collected from each participant and submitted for genetic analysis. Understanding the genetic predisposition to stroke could have major benefits for public health.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed by a study neurologist as having had a symptomatic ischemic stroke in the past.
* Head Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) done within 7 days of symptom onset confirms absence of etiology other than ischemic stroke.
* Subject reports having at least one living sibling with a stroke.
* Subject is 18 years of age or older.

Exclusion Criteria:

* The index ischemic stroke occurred within 48 hours after a cardiovascular or cerebrovascular procedure.
* The index ischemic stroke occurred within 60 days after a non-traumatic subarachnoid hemorrhage.
* The subject has brain biopsy-proven central nervous system vasculitis.
* The subject is known to have any one of the following genetic disorders: CADASIL (Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy), Fabry's disease, homocystinuria, MELAS (Mitochondrial myopathy, Encephalopathy, Lactic Acidosis, Stroke), or sickle cell anemia.
* The subject has a mechanical aortic valve or mechanical mitral valve.
* The subject had untreated or actively treated bacterial endocarditis at the time of the index ischemic stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in-patient or out-patient clinics, local community
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2000-12; Primary Completion 2009-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. Meschia, M.D., Principal Investigator — Mayo Clinic
Locations (32):
- United States (30):
  - University of South Alabama, Mobile, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - East Bay Region Assoc., Berkeley, California
  - Scripps Clinic, La Jolla, California
  - University of California, Davis, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Shands Jacksonville, Jacksonville, Florida
  - Mayo Clinic College of Medicine Jacksonville, Jacksonville, Florida
  - Florida Neurovascular Institute, Tampa, Florida
  - Cleveland Clinic - Florida, Weston, Florida
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Indiana University/Clarian Health Partners, Indianapolis, Indiana
  - Mercy Medical Center, Sioux City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rochester General Hospital, Rochester, New York
  - Helen Hayes Hospital, West Haverstraw, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Metro Health, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Penn. Med. Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Luther Midelfort Clinic, Eau Claire, Wisconsin
  - University of Wisconsin, Madison, Madison, Wisconsin
  - Froedtert Memorial Lutheran, Milwaukee, Wisconsin
- Canada (2):
  - Hospital Charles Le Moyne, Greenfield Park, Quebec
  - L'Enfant-Jesus Hospital, Québec, Quebec